CLINICAL TRIAL: NCT01458418
Title: A Trial of Montelukast for Maintenance Therapy of Eosinophilic Esophagitis in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to complete enrollment due to difficulty in finding subjects
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMH 11 01-007
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophil; Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Montelukast 10 mg/day (Experimental): Subjects will receive two 5mg tablets of Montelukast/day.
  Interventions: Drug: Montelukast
- Montelukast 5mg/day (Experimental): Subjects will receive one 5mg tablet of montelukast and 1 placebo tablet per day.
  Interventions: Drug: 5 mg Montelukast
- placebo (Placebo Comparator): Subjects will receive two placebo tablets per day.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Montelukast — Those in Montelukast 10mg/day group will receive two 5mg tablets of Montelukast.
  Other Names: Singulair
  Arms: Montelukast 10 mg/day
Other: placebo — Those in the placebo group will receive 2 placebo tablets per day. Those in the Montelukast 5mg/day will receive 1 placebo tablet per day.
  Arms: placebo
Drug: 5 mg Montelukast — Subject will receive one 5mg tablet of Montelukast and one placebo tablet per day.
  Other Names: Singulair
  Arms: Montelukast 5mg/day

SUMMARY:
Eosinophilic Esophagitis (EE) is a condition where eosinophils (a cell that fights infection) travel to the esophagus (the tube through which food passes to the stomach). These cells do not belong there and can cause pain, soreness, difficulty swallowing and sometimes vomiting.

Ways to treat this condition include medicine, not eating some foods, and drinking a specific formula (like milk) without eating any other foods. Doing these things can help fight off EE but these problems can come back when treatment is stopped. If EE symptoms go on for a long time, it can lead to the esophagus becoming narrow and feeling tight when eating and swallowing and surgery may be needed to widen the narrowed area to relieve the sensation of tightening.

Montelukast is a medicine that fights off a type of chemical that can be a magnet for eosinophils. People usually take this medicine to help treat their asthma. It is not approved to treat EE. This medication is taken once a day.

The purpose of this study is to see if Montelukast, compared to placebo, will help reduce the number of eosinophils in children with EE and help stop the tightening of the esophagus.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EE) is a disease diagnosed using both clinical and pathologic results. Presentation varies among age groups with younger children suffering from vomiting, failure to thrive, or food refusal and adolescents suffering from dysphagia, odynophagia, or food impaction. It is more prevalent in males. EE is suggested when an upper endoscopy yields eosinophils greater than 15 per high power field (hpf) in both the middle and distal esophagus. Therapy for EE depends upon age and ability to be compliant. Three main categories of treatment are options for families, including the use of medicines, removal of the most allergenic foods, and the use of an elemental diet (formula) (1-2). Treatment can be different within the two main phases of therapy for EE, initial and maintenance therapy. Initial therapy occurs when the patient is first diagnosed and has eosinophils over 15 per hpf and can last for years if the patient does not respond to treatment. Maintenance therapy only occurs after the patient has responded to treatment with a reduction of his/her eosinophil counts below 5 per hpf. Typically, medicinal therapy with steroids (either oral prednisone or swallowed fluticasone) improves eosinophil counts but has a large side effect profile suggesting that steroids are not ideal for maintenance therapy. Dietary therapies are effective in both treatment phases but many patients find it difficult to remain compliant with food restriction for a prolonged length of time. Unfortunately, EE recurs upon withdrawal of oral therapy (3-7).

EE is believed to be an imbalance of the TH1/TH2 immune system and is more prevalent in patients with asthma and allergies (8-9). Some EE centers have started treating patients with targeted elimination diets and elemental diets and are having good success. Unfortunately, most families and in particular teenagers, are noncompliant with the dietary therapies. Formula for the elemental diet is not covered by most insurance and is very costly as well. Therefore, finding a drug that would keep a patient with EE in maintenance therapy and reduce both the long term consequences of steroids and potential for esophageal strictures would be ideal.

Many adults with EE present with dysphagia or food impactions and subsequently are found to have an esophageal stricture requiring multiple esophageal dilatations for treatment. Esophageal subepithelial fibrosis has been found in the adult literature in patients with EE. Chehade et al evaluated distal esophageal biopsy specimens in children with EE, eosinophilic gastroenteritis, gastroesophageal reflux disease, and controls for the presence of increased collagen deposition indicative of fibrosis. They found that fibrosis was present in 57% of patients with EE, of which 42% had symptoms of dysphagia and 80% had food impactions. The degree of fibrosis was not associated with eosinophil count but was associated with eosinophilic degranulation (10). Upon degranulation, eosinophils release major basic protein (MBP) and transforming growth factor (TGF-β). MBP changes smooth muscle contractility by blocking M2 muscarinic receptors therefore changing the motility of the esophagus. TGF-β is believed to cause an increase in the production of the extracellular matrix and smooth muscle hypertrophy and hyperplasia leading to esophageal thickening and fibrosis. TGF-β is a key growth factor that increases fibroblasts and subsequent fibrosis in the lung as well. Corticosteroids have been shown to reverse esophageal remodeling, but no large clinical trials have evaluated the treatment of esophageal fibrosis related to EE. To quote Aceves and Ackerman: "[f]ibrosis likely contributes to multiple clinical aspects of EE, including dysphagia symptoms, disease chronicity, and stricture formation." Fibrosis is measured in esophageal tissue by evaluating the amount of collagen that is deposited. Trichrome stains specifically for collagen (11).

Patients with EE have an abundance of inappropriate cells within the esophagus, including eosinophils and mast cells. A normal esophagus is devoid of eosinophils. Mast cells likely have an active role in the development of eosinophilic esophagitis; unfortunately the precise mechanism is unknown. Mast cells are found in the majority of vascularized tissues and are abundant in the gastrointestinal tract. They are located in the submucosa and lamina propria. Within the esophagus specifically, they are found in the mucosa and submucosa with rare expansion into muscularis layer. With severe eosinophilic inflammation, mast cells can be seen in the muscularis layer. Biopsies from patients with EE have demonstrated marked increase in mast cells in the mucosal layer of the esophagus. There has been correlation of mast cell number with degree of eosinophilia. Mast cells within the GI tract contain tryptase as well as other preformed mediators and can synthesize mediators that promote inflammation. Tryptase may activate eosinophils and therefore induce eosinophilic degranulation and cytokine secretion. Mast cells release chemokines and leukotrienes specific to eosinophil recruitment. Ultimately mast cell mediators worsen edema, create more inflammation, induce smooth muscle contractility and potentially affect tissue fibrosis. Therefore, active mast cells are proinflammatory, modify esophageal function, and encourage the development of strictures (12). Mast cells may be a key component in the propagation of the inflammatory state as well as of significant importance in the development of fibrosis. Evaluating tryptase levels could lead to a better understanding of the inflammatory process and ultimate problem of fibrosis.

Eosinophils and mast cells contain leukotrienes in abundance. Cysteinyl leukotrienes are inflammatory mediators derived from arachidonic acid. They are important in eosinophil attraction and migration, smooth muscle bronchoconstriction, vascular permeability, and mucus hypersecretion (13). Montelukast is a leukotriene receptor antagonist and blocks specifically the leukotriene D4 (LTD4) receptor. Attwood et al treated 8 patients with EE with Montelukast for which 6 reported complete subjective improvement and 5 remained asymptomatic on a maintenance regimen. Treatment with Montelukast did not change the density of eosinophils present in the esophagus however (14). Montelukast has been used in mouse models to decrease fibrosis occurring in both the liver and the lung. El-Swefy and Hassanen performed a randomized study in which they subjected mice to one of 4 groups, no bile duct ligation plus saline, no bile duct ligation plus montelukast, bile duct ligation plus montelukast and bile duct ligation plus saline. Bile duct ligation induced inflammation leading to cirrhosis and fibrosis. They found that bile duct ligation increased the amount of TGF-β, which correlated with the amount of fibrosis found. Of more import is that montelukast significantly reduced the amount of fibrosis as well as decreased the amount of TGF-β (15). Izumo, Kondo, and Nagai evaluated the use of montelukast in the prevention of pulmonary fibrosis after exposure to bleomycin. They found that mice given montelukast had significantly lower levels of TGF-β and fibrosis of the lung (16).

The investigator's research focus throughout fellowship included several retrospective studies in eosinophilic esophagitis. One of the investiagotor's studies evaluated the management of both initial and maintenance therapy for EE within our department. The investigator wanted to know what medicines the majority of pediatric gastroenterologists at the investigator's institution were using to treat EE and how often patients were being reevaluated by endoscopy. The investigator also wanted to evaluate the use of montelukast in the treatment of EE. The investigator reviewed 1500 charts of patients who had undergone upper endoscopy and had a result of "esophagitis." Patients were then selected by the presence of greater than or equal to 20 eosinophils per high power field in at least one biopsy location. Of the 1500 charts the investigator evaluated, only 88 patients fulfilled criteria for EE. The investigator discovered that there is not a consistent standard of care within their department for the initial and maintenance treatment of EE. Many different medicines are trialed initially and patients undergo esophageal biopsies at different time intervals, contrary to what is recommended. The primary group of 88 patients was then separated into 49 patients who reached maintenance therapy (defined by less than 5 eosinophils per high power field) and 39 patients who never experienced improvement in their eosinophil counts. Of the 49 who reached maintenance therapy, 30 patients were treated with montelukast and had follow up endoscopy. The investigator evaluated peak eosinophil counts pre and post treatment, and contrary to their hypothesis, those patients treated with 5mg of montelukast had lower post treatment eosinophil counts than those treated with higher doses (10 and 20mg). This raised the possibility that the packaging differences of the two main doses had an impact in treatment. The investigator considered the possibility that the lower dosage of montelukast is protective since 5mg tablets are chewable and would yield a topical effect on the esophagus whereas the 10mg tablets are swallowed, not chewed. In addition, the investigator evaluated how often EE recurred and discovered there was a high rate of histologic recurrence. Also interesting to the investigator was the lower recurrence rate in patients given 5mg of montelukast compared to 10mg and 20mg doses. These results were not expected and deserve further evaluation. If montelukast can prevent fibrosis through a topical effect, then its therapeutic potential is huge in the treatment of EE.

The investigator has developed a study that will investigate the use of montelukast in total vs placebo as well as allow them to look for dosing effects within montelukast in the treatment of eosinophilic esophagitis. The primary objective is to evaluate if montelukast will keep eosinophil counts low enough for the patient to remain in remission and if so, is there a particular dose of montelukast that will achieve this in a greater proportion. All patients will be maintained on a proton pump inhibitor (PPI) at baseline so that patients receiving placebo will still receive standard of care treatment. Many GI practitioners at this institution will place patients with EE on montelukast as part of standard of care treatment at varying doses without any good literature to support this use. The investigator's goal is to determine if montelukast is a valuable therapy in the treatment of EE. The investigator's study will also evaluate histological stains that may show an improvement with the use of montelukast, even if the eosinophil counts do not change, as the chemicals released by eosinophils and mast cells may be of primary import in the continuation of EE.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 2-17
* Presence of more than 15 eosinophils per hpf on original endoscopy and less than 5 eosinophils/hpf on the most recent endoscopy
* Concurrent PPI for 1 month at 1-2mg/kg/dose prior to endoscopy or have a negative pH study
* English speaking
* Ability to undergo a follow up endoscopy between 12 and 13 weeks after the start of the study
* Procurement of written informed consent signed by the subject's legal guardian and study investigator (s) and subject assent.

Exclusion Criteria:

* Subjects with eosinophils in stomach and duodenum on original endoscopy.
* Subjects requiring oral prednisone within 1 month of current endoscopy.
* Subjects with diagnosis of other co-morbid diseases such as heart disease, renal disease, autoimmune disease, an immunodeficiency, diabetes, phenylketonuria, or thyroid disease.
* Subjects using Montelukast within one month of current endoscopy
* Subjects with concurrent use of phenobarbital or rifampin

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Page, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Rothenberg ME. Biology and treatment of eosinophilic esophagitis. Gastroenterology. 2009 Oct;137(4):1238-49. doi: 10.1053/j.gastro.2009.07.007. Epub 2009 Aug 15. PMID 19596009
- [Background] Konikoff MR, Noel RJ, Blanchard C, Kirby C, Jameson SC, Buckmeier BK, Akers R, Cohen MB, Collins MH, Assa'ad AH, Aceves SS, Putnam PE, Rothenberg ME. A randomized, double-blind, placebo-controlled trial of fluticasone propionate for pediatric eosinophilic esophagitis. Gastroenterology. 2006 Nov;131(5):1381-91. doi: 10.1053/j.gastro.2006.08.033. Epub 2006 Aug 16. PMID 17101314
- [Background] Schaefer ET, Fitzgerald JF, Molleston JP, Croffie JM, Pfefferkorn MD, Corkins MR, Lim JD, Steiner SJ, Gupta SK. Comparison of oral prednisone and topical fluticasone in the treatment of eosinophilic esophagitis: a randomized trial in children. Clin Gastroenterol Hepatol. 2008 Feb;6(2):165-73. doi: 10.1016/j.cgh.2007.11.008. PMID 18237866
- [Background] Dohil R, Newbury R, Fox L, Bastian J, Aceves S. Oral viscous budesonide is effective in children with eosinophilic esophagitis in a randomized, placebo-controlled trial. Gastroenterology. 2010 Aug;139(2):418-29. doi: 10.1053/j.gastro.2010.05.001. Epub 2010 May 7. PMID 20457157
- [Background] Markowitz JE, Spergel JM, Ruchelli E, Liacouras CA. Elemental diet is an effective treatment for eosinophilic esophagitis in children and adolescents. Am J Gastroenterol. 2003 Apr;98(4):777-82. doi: 10.1111/j.1572-0241.2003.07390.x. PMID 12738455
- [Background] Assa'ad AH, Putnam PE, Collins MH, Akers RM, Jameson SC, Kirby CL, Buckmeier BK, Bullock JZ, Collier AR, Konikoff MR, Noel RJ, Guajardo JR, Rothenberg ME. Pediatric patients with eosinophilic esophagitis: an 8-year follow-up. J Allergy Clin Immunol. 2007 Mar;119(3):731-8. doi: 10.1016/j.jaci.2006.10.044. Epub 2007 Jan 25. PMID 17258309
- [Background] Blanchard C, Wang N, Rothenberg ME. Eosinophilic esophagitis: pathogenesis, genetics, and therapy. J Allergy Clin Immunol. 2006 Nov;118(5):1054-9. doi: 10.1016/j.jaci.2006.07.038. Epub 2006 Sep 18. PMID 17088129
- [Background] Blanchard C, Rothenberg ME. Basic pathogenesis of eosinophilic esophagitis. Gastrointest Endosc Clin N Am. 2008 Jan;18(1):133-43; x. doi: 10.1016/j.giec.2007.09.016. PMID 18061107
- [Background] Chehade M, Sampson HA, Morotti RA, Magid MS. Esophageal subepithelial fibrosis in children with eosinophilic esophagitis. J Pediatr Gastroenterol Nutr. 2007 Sep;45(3):319-28. doi: 10.1097/MPG.0b013e31806ab384. PMID 17873744
- [Background] Aceves SS, Ackerman SJ. Relationships between eosinophilic inflammation, tissue remodeling, and fibrosis in eosinophilic esophagitis. Immunol Allergy Clin North Am. 2009 Feb;29(1):197-211, xiii-xiv. doi: 10.1016/j.iac.2008.10.003. PMID 19141355
- [Background] Wershil BK. Exploring the role of mast cells in eosinophilic esophagitis. Immunol Allergy Clin North Am. 2009 Feb;29(1):189-95, xiii. doi: 10.1016/j.iac.2008.09.006. PMID 19141354
- [Background] Lucendo AJ, Bellon T, Lucendo B. The role of mast cells in eosinophilic esophagitis. Pediatr Allergy Immunol. 2009 Sep;20(6):512-8. doi: 10.1111/j.1399-3038.2008.00798.x. Epub 2008 Aug 4. PMID 18681944
- [Background] Attwood SE, Lewis CJ, Bronder CS, Morris CD, Armstrong GR, Whittam J. Eosinophilic oesophagitis: a novel treatment using Montelukast. Gut. 2003 Feb;52(2):181-5. doi: 10.1136/gut.52.2.181. PMID 12524397
- [Background] El-Swefy S, Hassanen SI. Improvement of hepatic fibrosis by leukotriene inhibition in cholestatic rats. Ann Hepatol. 2009 Jan-Mar;8(1):41-9. PMID 19221533
- [Background] Izumo T, Kondo M, Nagai A. Cysteinyl-leukotriene 1 receptor antagonist attenuates bleomycin-induced pulmonary fibrosis in mice. Life Sci. 2007 Apr 24;80(20):1882-6. doi: 10.1016/j.lfs.2007.02.038. Epub 2007 Mar 12. PMID 17397875
- [Background] Montagna NA, de Oliveira ML, Mandarim-de-Lacerda CA, Chimelli L. Leprosy: contribution of mast cells to epineurial collagenization. Clin Neuropathol. 2005 Nov-Dec;24(6):284-90. PMID 16320824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place between 9/17/2012 and 1/7/2013 in a clinical setting.
Pre-assignment Details: There were no pre-assignment details. All inclusion/exclusion criteria were measured using existing, standard of care data. All subjects who signed informed consent were randomized (although it is not now know which arm they were randomized to as no unblinding was ever done due to low enrollment and lack of data).
Groups:
- Subjects Who Were Not Unblinded so Arm is Unknown: Subjects were never unblinded and no results were reported due to small number of enrolled subjects and lack of amount of data to show any demonstrable differences.
Period: Overall Study
Arm/Group | Montelukast 10 mg/Day | Montelukast 5mg/Day | Placebo | Subjects Who Were Not Unblinded so Arm is Unknown
Started | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were never unblinded as study was stopped prior to data analysis (number of subjects too low to create generalizable knowledge)
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 10 mg/Day | Montelukast 5mg/Day | Placebo | Subjects Who Were Not Unblinded so Arm is Unknown | Total
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 4 | 4
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  |  |  | 10 [5 to 15] | 10 [5 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 2
  Male | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States |  |  |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Eosinophil Count
Description: Eosinophils/high powered field(hpf) in the mid esophagus will be measured after 12 weeks of therapy.
Time Frame: 12 weeks
Population: Subjects were not unblinded due to inability to enroll numbers to create generalizable knowledge, so we don't know how many subjects were in each arm.
Measure: Mean (Full Range); unit: Eosinophils/HPF
Groups:
- Subjects Whose Arm is Unknown Due to Not Being Unblinded: subjects were never unblinded as data was never analyzed due to too few subjects to create generalizable knowledge.
Arm/Group | Montelukast 10 mg/Day | Montelukast 5mg/Day | Placebo | Subjects Whose Arm is Unknown Due to Not Being Unblinded
Number analyzed (Participants) | 0 | 0 | 0 | 4
Eosinophils/HPF |  |  |  | 8 [2 to 20]

ADVERSE EVENTS:
Time Frame: 14 weeks. From time of enrollment to completion of last study visit.
Arm/Group | Montelukast 10 mg/Day | Montelukast 5mg/Day | Placebo | Subjects Who Were Not Unblinded so Arm is Unknown
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
Study was difficult to enroll for and study was stopped due to length of time it took to enroll and sponsor pulling funding prior to enrollment meeting goal to have generalizable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No